CLINICAL TRIAL: NCT07119437
Title: Low Impact Laparoscopy In Bariatric Surgery- A Monocentric Randomised Trial Comparing Low-Pressure Pneumoperitoneum Plus Microsurgery Versus Standard Laparoscopy
Brief Title: Low Impact Laparoscopy In Bariatric Surgery
Acronym: LILYBET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 251.24 CET2 cbm
Record Dates: First submitted 2025-02-10; First posted 2025-08-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Morbid
Keywords: obesity; low impact laparoscopy; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Microsurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Pneumoperitoneum Laparoscopy with microsurgery (Experimental)
  Interventions: Procedure: low pneumoperitoneum laparoscopy with microsurgery
- standard laparoscopy (Active Comparator)
  Interventions: Procedure: standard laparoscopy

INTERVENTIONS:
Procedure: low pneumoperitoneum laparoscopy with microsurgery — Use of low pressure for pneumoperitoneum (8-10 mmHg) and mini surgical access for bariatric procedure (sleeve gastrectomy).
  Arms: Low Pneumoperitoneum Laparoscopy with microsurgery
Procedure: standard laparoscopy — Standard laparoscopy (12-14 mmHg) and normal surgical access for bariatric procedures (sleeve gastrectomy).
  Arms: standard laparoscopy

SUMMARY:
The goal of this clinical trial is to learn if low pressure pneumoperitoneum and small incisions (low impact laparoscopy, LIL) works to reduce pain and improve pulmonary function in patients underwent to bariatric surgery.

It will also learn about the safety and patients' satisfaction of the procedure. The main questions it aims to answer are:

Does LIL lower post surgical pain and improve pulmonary function? Is LIL safe for obese patients? Researchers will compare LIL to standard laparoscopy performing sleeve gastrectomy in patients with obesity.

Participants will:

be randomised to LIL group or standard laparoscopy. After the operation the researchers will evaluate the pain and the efficiency of lung ventilation at pre-established intervals. after 3 months the patients will complete a questionnaire on aesthetic satisfaction and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years-old and 65 years-old
* BMI (Body Mass Index) >35 Kg/m2 and < 45 Kg/m2;
* Patients candidate to sleeve gastrectomy

Exclusion Criteria:

* Patients with neurological and/or psychiatric disorders
* Patients with Chronic Pain Syndrome
* Patients with a history of surgical procedures using a laparotomic approach in the upper abdominal quadrants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
POST OPERATIVE PAIN | FROM THE ENTER IN PACU TO 36 HOURS POST- SURGERY
  Post-operative pain (AS REST PAIN AND MOVIMENT PAIN) will be assessed using the Numeric Pain Rating Scale (NRS), which rates pain from 0 to 10. 0 is defined as no pain, while 10 represents the maximum pain.
  0 is the best result, 10 the worst. The questionnaire will be administered in the PACU and at 6, 12, 24, and 36 hours after the end of the procedure.
Pulmonary performance | from surgery to 24 hours post-surgery
  Efficiency of ventilation will be evaluated recording the values of Maximum Inspiratory Pressure (MIP), maximum expiratory pressure (MEP), Peak expiratory flow (PEF)

SECONDARY OUTCOMES:
USE OF Analgesics | from surgery to 36 hours post-surgery
  Comparison of analgesic use between the two groups during post-operative recovery
operative time | from the surgical incision to the last skin stitch
  Comparison of opertive time between the two groups
Rate of conversion to standard laparoscopy | from the beginning of surgery to the end of surgery
  Record the number of cases in the operative group where conversion to a standard laparoscopic approach was necessary, with pressure values > 10 mmHg for more than 20% of the duration of the procedure. Also analyzing the results for BMI subgroups.
Rate of laparotomy conversion | from the beginning of surgery to the end of surgery
  Number of cases in which the surgical procedure had to be converted from laparoscopy to an open approach.
Ambulation Time | From the end of surgery up to 24 hours post-surgery
  Comparison of mobilization time between the two groups
The time to first flatus | From the end of surgery up to 48 hours post-surgery
  Compare the time to intestinal motility recovery between the two groups.
Liver Function | first and second post-operative day
  Comparison between the two groups of liver function tests that include alanine transaminase (ALT, Normal values 0-55 U/L) , aspartate transaminase (AST, normal values 5-34 U/L), alkaline phosphatase (ALP normal values 53-141 U/L) and gamma-glutamyl transferase (GGT, normal values 8-33 U/L).
Post-operative hospital stay | from the day of surgery up to 30 days
  Post-operative hospital stay
Postoperative complications | from surgery to 30 days after surgery
  All postoperative complications
First Operator Comfort | during surgery
  Evaluate the comfort of the operating surgeon related to the adequate exposure of the surgical field during the procedure using a 5-point surgical rating scale for laparoscopic surgical workspace. The scale ranges from 1 to 5, where 1 corresponds to the worst possible outcome, while 5 represents the best possible outcome.
Aesthetic satisfaction | from surgery to 3-month post surgery
  Evaluate the degree of aesthetic and overall satisfaction of patients by administering to them, 3 months after the intervention, the Patient Scar Assessment Scale (PSAS), a validated tool for scar assessment, and the Ultimate Question (UQ), related to overall satisfaction.
  These tests are administered together and the patient, who responds to 8 different items, assigning a score from 1 to 10. The maximum test score is 80, indicating the highest satisfaction, while the minimum score is 8, corresponding to the worst possible outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Campus Bio-Medico, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided